CLINICAL TRIAL: NCT07315113
Title: A Phase 1b Clinical Study of NXP900 in Combination With Osimertinib in Subjects With Advanced, EGFRMut+ Non-Small Cell Lung Cancer
Brief Title: Study of NXP900 With Osimertinib in Subjects With Advanced, EGFR-Mutated Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nuvectis Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NXP900-103
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: EGFR Mutation Positive Non-small Cell Lung Cancer; EGFR Mutated Non-small Cell Lung Cancer Patients
Keywords: EGFR; Epidermal growth factor receptor; NSCLC; non-small cell lung cancer; lung cancer; osimertinib; NXP900; EGFR mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Exploration (Part 1) (Experimental): Escalating doses of NXP900 given with osimertinib
  Interventions: Drug: NXP900; Drug: Osimertinib

INTERVENTIONS:
Drug: NXP900 — NXP900 is an orally administered inhibitor of SRC family kinases (SFK)
Drug: Osimertinib — Osimertinib is an orally available, irreversible, mutant-selective, epidermal growth factor receptor (EGFR) inhibitor

SUMMARY:
This is a multi-center, open label, Phase 1b study of NXP900 in combination with osimertinib in subjects with advanced, progressing, EGFR-mutated non-small cell lung cancer (NSCLC)

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. 18 years old or older.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Unresectable, metastatic or locally advanced EGFR-mutated NSCLC.
5. Prior treatment with osimertinib as first or second line, as single agent or in combination with chemotherapy, in the metastatic or locally advanced setting.

Exclusion Criteria:

1. Subject's cancer has a known oncogenic driver alteration other than EGFR.
2. Known EGFR mutations that cause resistance to osimertinib
3. Known human epidermal growth factor receptor 2 (HER2) overexpression
4. Any contraindications to treatment with osimertinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment related adverse events and/or clinical laboratory abnormalities | Up to 30 days post treatment
Objective response rate (ORR) | Up to approximately 12 months
  Best response of complete response (CR) or partial response (PR) per RECIST 1.1
Duration of Response (DoR) | Up to approximately 12 months
  Confirmed CR or PR from the first documented response to the date of documented disease progression or death.
Disease Control Rate (DCR) | Up to approximately 12 months
  The proportion of patients with stable disease (SD), partial response (PR), or complete response (CR).

CONTACTS AND LOCATIONS:
Overall Officials: Zofia Piotrowska, MD, MHS, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - NEXT Houston, Houston, Texas
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No